CLINICAL TRIAL: NCT06829134
Title: Clinical Analysis of the Antihypertensive Effect of Laparoscopic Peripheral Nerve Blockade of the Renal Artery in Patients With Retroperitoneal Disease and Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-489
Record Dates: First submitted 2025-01-22; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Retroperitoneal Disease
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will undergo surgery related to the primary disease in addition to laparoscopic renal artery perivascular nerve blockade.
  Interventions: Procedure: laparoscopic renal artery perivascular nerve blockade; Procedure: surgery related to the primary disease
- control group (Sham Comparator): The control group will only receive surgery related to the primary disease. Such as laparoscopic partial nephrectomy, laparoscopic adrenalectomy etc.
  Interventions: Procedure: surgery related to the primary disease

INTERVENTIONS:
Procedure: laparoscopic renal artery perivascular nerve blockade — 1. When only the main renal artery is present: The complete dissection of the renal artery should be performed in the distal 2/3 portion, close to the renal hilum. The connective tissue and nerve tissue within a 1 cm radius from the center of the renal artery lumen must be completely separated (using instruments such as an ultrasonic scalpel or monopolar hook, etc.). The length of the dissected renal artery should be at least 0.5 cm, forming a dissection ring.
  2. When accessory renal arteries are present: In addition to the main renal artery meeting the aforementioned standards, the accessory renal arteries must also be dissected. The radius of the dissection ring should be 0.7 cm, with a length ranging from 0.3 to 0.5 cm.
  3. When renal polar arteries are present: Dissection may be performed appropriately based on the surgical conditions.
  4. The prerequisite is to ensure the safety of the surgery, specifically the safe resection of the primary lesion.
  Arms: experimental group
Procedure: surgery related to the primary disease — The surgeries related to the primary disease include laparoscopic partial nephrectomy, laparoscopic adrenalectomy, and other similar procedures.

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of laparoscopic renal artery nerve blockade surgery in patients with retroperitoneal diseases complicated by hypertension.

The study aims to address the following two questions:

1. Can laparoscopic renal artery perivascular nerve blockade reduce postoperative blood pressure and decrease the dependence on antihypertensive medications in patients with retroperitoneal diseases and hypertension?
2. What is the safety profile of the procedure, and does it lead to any complications?

The researchers will randomly assign patients to the experimental group and the control group. The experimental group will undergo surgery related to the primary disease in addition to laparoscopic renal artery perivascular nerve blockade, while the control group will only receive surgery related to the primary disease. This design allows for a comparison of the effects of renal artery perivascular nerve blockade on postoperative blood pressure.

Participants will:

1. Patients will undergo either surgery related to the primary disease combined with renal artery perivascular nerve blockade, or surgery related to the primary disease alone.
2. For the three months following surgery, the antihypertensive medication regimen will remain unchanged from the preoperative plan. At the end of the three-month period, patients will visit the hospital for 24-hour ambulatory blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Renal artery diameter ≥ 4 mm, length ≥ 20 mm.
* Age between 18 and 75 years, male or female.
* Scheduled to undergo laparoscopic surgery: The patient has a clear diagnosis of adrenal tumor, early-stage renal malignancy, renal cyst, etc., and meets the surgical indications recommended by guidelines or relative surgical indications but has a strong willingness for surgery. The patient requires surgery (such as laparoscopic partial adrenalectomy, laparoscopic unilateral adrenalectomy, laparoscopic partial nephrectomy, laparoscopic renal cyst decapitation, etc.) and meets the surgical conditions.
* A clear diagnosis of hypertension: Either the patient has never used antihypertensive medications, with in-office blood pressure ≥ 140/90 mmHg and < 180/110 mmHg, or 24-hour daytime ambulatory blood pressure ≥ 135/85 mmHg and < 170/105 mmHg. Alternatively, the patient has been diagnosed with hypertension and has been taking antihypertensive medications for at least 4 weeks.
* Estimated glomerular filtration rate (eGFR) ≥ 45 ml/min/1.73 m².
* The patient is willing and able to comply with the study protocol, provide written informed consent, and agrees to participate in follow-up assessments.

Exclusion Criteria:

* Renal artery abnormalities: Hemodynamic or anatomical stenosis (≥50%) of one renal artery; post-renal artery balloon angioplasty or stent placement;
* Cardiovascular risk factors: Including myocardial infarction, unstable angina, or cerebrovascular events within the past 6 months; extensive atherosclerosis with intravascular thrombosis or unstable plaques; and significant hemodynamic changes due to heart valve disease;
* History of similar surgeries: Such as previous renal sympathetic nerve ablation via catheter;
* Other severe organic diseases;
* Participation in other clinical studies;
* Investigator's judgment: The investigator determines that, based on medical expertise, the patient is unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The blood pressure values at 3 months post-surgery. | 3 months
  The average systolic blood pressure (ASBP) during 24-hour ambulatory blood pressure monitoring at 3 months post-surgery.

SECONDARY OUTCOMES:
The blood pressure values at other different time points. | 1 month, 3 months，6 months, 12 months, and 24 months
  The 24-hour ambulatory blood pressure data at 1 month, 6 months, 12 months, and 24 months post-surgery, as well as the dynamic blood pressure data at 3 months post-surgery, excluding the primary outcomes.
antihypertensive medications | 1 month, 3 months，6 months, 12 months, and 24 months
  The use of antihypertensive medications at 1 month, 3 months, 6 months, 12 months, and 24 months post-surgery.
Health status. | 1 month, 3 months，6 months, 12 months, and 24 months
  At each time point, health status will be assessed and quantified using the EuroQoL Five-Dimensions Three-Level (EQ-5D-3L) standardized scale.
Pain score | 1 month, 3 months，6 months, 12 months, and 24 months
  At each time point, Pain scores will be assessed and quantified using the Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No